CLINICAL TRIAL: NCT05081713
Title: Locomotor Recovery and Compensation Post-stroke (LRC)
Acronym: LRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Rehabilitation Hospital of Indiana (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, George Hornby, Professor of Physical Medicine, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IU2011618233; 1R01NS118009 (NIH)
Record Dates: First submitted 2021-09-24; First posted 2021-10-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: two separate longitudinal observational studies with interventions at different phases (duration) of recovery post-stroke
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Other): Observational evaluations for 6 months followed by 3-4 months of high-intensity training (HIT)
  Interventions: Behavioral: high-intensity training focused on stepping in variable contexts
- Phase 2 (Other): Observational evaluations for 1 month followed by 3-4 months of high-intensity training (HIT)
  Interventions: Behavioral: high-intensity training focused on stepping in variable contexts

INTERVENTIONS:
Behavioral: high-intensity training focused on stepping in variable contexts — Approximately 10 weeks (~30 sessions) of high-intensity training
  Other Names: HIT

SUMMARY:
The proposed research will characterize of the time course of neurological and locomotor recovery as well as development of compensatory strategies throughout sub-acute and chronic phases post stroke. In addition, we will also investigate the extent to which measures of recovery and compensation are malleable and can be altered with specific interventions in both the early and late stages post-stroke. Delineation of the time course of development and magnitude of patterns of recovery and compensation should result in alternative predictive "rules' regarding how patients early post-stroke could recovery functional and neurological function.

DETAILED DESCRIPTION:
Recovery of locomotion is a primary goal of rehabilitation post-stroke and a major determinant of future morbidity and mortality. While substantial recovery is observed early post-stroke, recent evidence suggests the magnitude and time course of recovery is deterministic and based primarily on initial motor deficits. The "proportional recovery" rule suggests ~70% of neurological recovery (measured by the lower limb Fugl-Meyer Assessment - LL-FMA) is typically achieved and is not influenced by the dosage of therapy. These findings suggest the physical interventions applied to patients are of minimal importance to long-term recovery. That hypothesis conflicts directly with our recent efforts suggesting that maximizing the amount and intensity of task-specific (stepping) practice (high-intensity training; HIT) directly influences gains in locomotor function. Providing HIT at heart rates (HRs) greater than traditional aerobic paradigms (mean 110% baseline HRmax) is associated with gains in locomotor speed, which challenges the notion of "proportional recovery".

These conflicting hypotheses likely arise from differences in terminology and methodology used to characterize recovery post-stroke. First, the traditional measure of neurological recovery (LL-FMA) does not adequately characterize other impairments (strength, postural stability) that are more closely associated to locomotor function and are responsive to physical interventions. Second, despite gains in selected impairments, patients often utilize alternative (compensatory) movement patterns to accomplish locomotor tasks. More directly, locomotor recovery (i.e., speed/distance) is often accomplished using strategies employed prior to stroke and compensatory strategies, particularly in those with substantial impairments.

Our central hypothesis is that if changes in neurological recovery are deterministic, other measures of locomotor recovery or compensations may also be predictable. Our published data detail how HIT or conventional interventions can alter impairments and locomotor recovery, as well as changes in locomotor compensations. More directly, our data provide evidence that specific subgroups of patients demonstrate substantial compensations with improved recovery, whereas others reveal limited changes despite similar interventions. Data that detail the progression of neurological recovery, locomotor recovery, and locomotor compensations throughout the subacute to chronic phase post-stroke and their responsiveness to HIT is uncertain. Similar to upper limb recovery algorithms, predictions of mobility outcomes could provide valuable information to clinicians who make decisions regarding patient's prognosis, including whether patients will be able to walk with or without assistance or at certain speeds, and what compensatory strategies they may require to ambulate independently (braces, devices or altered movement patterns). The overarching goal of this project is to examine the time course of neurological and locomotor recovery, and associated compensatory strategies, over the subacute to chronic stages post-stroke and their responsiveness to HIT.

ELIGIBILITY:
Inclusion criteria:

* individuals early post-stroke (<15-30 days)
* first ever stroke
* unilateral hemiparesis
* currently receiving inpatient rehabilitation
* ability to follow 1-step commands
* provision of informed consent
* medical clearance from the rehabilitation physician to participate. \

Exclusion criteria:

* uncontrolled cardiovascular, metabolic or respiratory disease that limits exercise participation (e.g., congestive heart failure, resting blood pressure > 200/110 mmHg, uncontrolled diabetes, end-stage renal disease)
* absolute criteria for termination of exercise testing during initial and repeated ECG testing during graded exercise testing using ACSM guidelines .
* other orthopedic or neurological disorder that limited walking prior to stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Gait speed | 15 days post-stroke
  Walking speed over 6 m
Gait speed | 1 month
  Walking speed over 6 m
Gait speed | 2 months,
  Walking speed over 6 m
Gait speed | 4 months,
  Walking speed over 6 m
Gait speed | 6 months,
  Walking speed over 6 m
Gait speed | 9 months,
  Walking speed over 6 m
Gait speed | 12 months
  Walking speed over 6 m
Walking distance | 15 days post-stroke,
  Distance covered over 6 min
Walking distance | 1 month,
  Distance covered over 6 min
Walking distance | 2 months,
  Distance covered over 6 min
Walking distance | 4 months,
  Distance covered over 6 min
Walking distance | 6 months,
  Distance covered over 6 min
Walking distance | 9 months,
  Distance covered over 6 min
Walking distance | 12 months
  Distance covered over 6 min

SECONDARY OUTCOMES:
peak knee angle | 6 months
  peak knee angle during swing phase

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after completion of study for 3 years